CLINICAL TRIAL: NCT00893386
Title: Attain StarFix® Model 4195 LV Lead Extraction Study
Brief Title: Attain StarFix® 4195 Lead Extraction Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: StarFix Extraction
Record Dates: First submitted 2009-04-28; First posted 2009-05-06 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure; Indications for Lead Removal
Keywords: Extraction; Removal; Lead; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-4195 Lead, 181 days: Patients with a Medtronic LV Lead, other than Model 4195, implanted at least 181 days
  Interventions: Procedure: LV Lead Extraction
- 4195 Lead, 181 days: Patients with a Medtronic Model 4195 LV Lead implanted at least 181 days
  Interventions: Procedure: LV Lead Extraction
- 4195 Lead, 90-180 days: Patients with Medtronic Model 4195 LV Lead implanted for 90-180 days
  Interventions: Procedure: LV Lead Extraction

INTERVENTIONS:
Procedure: LV Lead Extraction — Removal of a LV lead using any tools & techniques.

SUMMARY:
The purpose of this study is to characterize the removability of the Attain StarFix® Model 4195 Left Ventricular (LV) Lead (StarFix®). The goal of the trial is to evaluate the lead removal success in patients that are indicated for left ventricular lead removal. This study is required by the Food and Drug Administration (FDA) as a condition of approval for the Attain StarFix® Model 4195 LV Lead.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a Class I/II indication and/or physician discretion for left ventricular lead removal
* Medtronic Model 4195 LV lead implanted for at least 181 days at time of extraction, or other Medtronic LV Lead (non-Model 4195) implanted for at least 181 days at time of extraction, or Medtronic Model 4195 LV lead implanted for 90-180 days
* Intention to remove the LV lead prior to the extraction procedure
* Subject is 18 years of age or older
* Subject (or subject's legally authorized representative) has signed and dated the Patient Consent Form and is willing and able to comply with the protocol

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be chosen by investigators participating in the study at up to 25 experienced extraction centers throughout the United States and Canada. Patients of both genders that are indicated for a Model 4195 or a non-Model 4195 Medtronic lead extraction who meet all inclusion criteria may be in the study.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2009-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Removal success of LV leads implanted for more than 180 days | More than 180 days post-implant

SECONDARY OUTCOMES:
Success of lead removal by how long the lead has been implanted | More than 180 days post-implant
Adverse Events that are related to the LV lead, the extraction procedure, or the extraction tool. | 0 to 45 days post-lead extraction
Removal success of Medtronic Model 4195 LV Leads implanted for 90-180 days | 90 -180 days post-implant
Summary of tools & techniques used to remove LV leads. | More than 180 days post-implant

CONTACTS AND LOCATIONS:
Overall Officials: 4195 Extraction Study Team, Study Chair — Medtronic
Locations (24):
- United States (21):
  - Phoenix, Arizona
  - Burbank, California
  - Long Beach, California
  - Aurora, Colorado
  - Miami, Florida
  - Chicago, Illinois
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - Spokane, Washington
- Canada (3):
  - Ottawa, Ontario
  - Toronto, Ontario
  - Sainte-Foy, Quebec